CLINICAL TRIAL: NCT06508593
Title: Metabolomics Analysis of Acute Kidney Injury and Delirium After Cardiac Surgery: Single Center, Prospective, Observational Study
Brief Title: Metabolomics Analysis of Acute Kidney Injury and Delirium After Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Chong Lei, MD & phD, Principal investigator, Head of Anesthesia Clinical Research Center, Xijing Hospital, Xijing Hospital
Other Study IDs: KY20242228-C-1
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: AKI - Acute Kidney Injury; Delirium, Postoperative
Keywords: AKI; Delirium; Cardiac surgery; Metabolomics
MeSH Terms: conditions — Acute Kidney Injury; Emergence Delirium; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- AKI group: Patients developed AKI after cardiac surgery
  Interventions: Diagnostic Test: Serum metabolic profile
- Delirium group: Patients developed delirium 5 days after cardiac surgery
  Interventions: Diagnostic Test: Serum metabolic profile
- AKI and delirium group: Patients developed AKI and delirium after cardiac surgery
  Interventions: Diagnostic Test: Serum metabolic profile
- Control group: Patients didn't develope AKI or delirium after cardiac surgery
  Interventions: Diagnostic Test: Serum metabolic profile

INTERVENTIONS:
Diagnostic Test: Serum metabolic profile — Venous serum samples were analyzed for serum metabolic profiles using liquid chromatography-mass spectrometry (LC-MS) and gas chromatography-mass spectrometry (GC-MS) non targeted metabolomics techniques

SUMMARY:
Clinical evidence suggests that renal injury leads to changes in the structure of the cerebral cortex in patients, suggesting the existence of the renal brain axis. Therefore, some scholars have proposed that AKI may be an important cause of secondary injuries such as delirium. Approximately 60% of AKI patients in clinical practice experience delirium.Although the underlying mechanism associated with acute renal injury and delirium is still unclear, it has been recognized that it increases incidence rate and mortality, prolongs hospital stay, and accelerates long-term cognitive decline. The investigators assume that the serum metabolic profiles of patients with delirium and AKI after cardiac surgery, with delirium only, with AKI only, and without delirium or AKI after surgery can be compared separately to explore the mechanisms of complications and the interaction mechanisms between organ damage after extracorporeal circulation cardiac surgery, and to identify metabolic markers specific to complications, identify patients with increased susceptibility, and provide reference for early diagnosis of complications and basis for early intervention.

DETAILED DESCRIPTION:
Approximately 2 million patients undergo cardiac surgery every year, of which approximately 20% to 30% experience cardiac surgery related acute kidney injury (CSA-AKI). At least 3% of CSA-AKI patients require temporary renal replacement therapy, and approximately 25% of patients will develop chronic kidney disease2 in three years. Several retrospective cohort studies have reported a significant correlation between AKI related to cardiac surgery and subsequent occurrence of chronic kidney disease, end-stage renal disease, heart failure, and major cardiovascular adverse events. Meanwhile, the occurrence of CSA-AKI is significantly associated with higher hospitalization costs and increased short-term and long-term postoperative mortality rates, with 5-year and 7-year cohort survival rates of 54% and 38%, respectively.

The pathogenesis of CSA-AKI is complex, caused by various potential kidney damage during the perioperative period. The commonality of these injuries is that the oxygen delivery into the kidneys is lower than the oxygen demand of the kidneys, leading to renal tubular injury. Hypothetical mechanisms leading to CSA AKI include hypoperfusion 8, atherosclerotic embolism, toxic effect of nephrotoxin 9, inflammation and oxidative stress hypothesis 1, etc. The hemodynamic changes, reduced oxygen supply, inflammation, and oxidative stress caused by these mechanisms may all lead to AKI10. In view of the high incidence rate of CSA AKI and its potentially devastating sequelae, it is urgent for clinical staff to understand how to best prevent and mitigate CSA-AKI.

Due to special reasons such as large surgical trauma, high surgical stress, extracorporeal circulation, and the need to be transferred to the cardiovascular intensive care unit after surgery, the incidence of postoperative delirium in the heart and large blood vessels (PODOCVS) is as high as 26% to 52%. PODOCVS refers to an acute neurological disorder that occurs after surgery, mainly characterized by confusion in thinking, decreased spatial and temporal positioning abilities. Related studies suggest that PODOCVS significantly prolongs patients' mechanical ventilation time, ICU stay time, incidence of complications, and is closely related to long-term cognitive decline and increased long-term mortality. However, the mechanism research of PODOCVS is still in its initial stage. Existing research has shown that multiple factors such as surgical trauma, extracorporeal circulation, and intraoperative management work together to cause neural network dysfunction through various mechanisms and pathways, leading to the occurrence of PODOCVS. The neuroinflammation theory plays a crucial role in the pathogenesis of PODOCVS. Acute peripheral inflammation stimulation induces the expression of inflammatory factors (IL-6, IL-8, IL-1 β α, TNF - α) in the central nervous system, leading to neuronal synaptic dysfunction, hippocampal dependent memory damage, and subsequent behavioral and cognitive symptoms. Some scholars have also proposed that damage to the anatomical structure and functional abnormalities of the central nervous system are potential mechanisms of PODOCVS. Through head magnetic resonance imaging of 116 patients undergoing elective cardiac surgery, it was found that the decrease in gray matter volume may be related to delirium during surgery. PODOCVS has many adverse effects on patient prognosis, therefore its mechanism research is crucial for the correct prevention and management of PODOCVS.

Clinical evidence suggests that renal injury leads to changes in the structure of the cerebral cortex in patients, suggesting the existence of the renal brain axis. Therefore, some scholars have proposed that AKI may be an important cause of secondary injuries such as delirium. Approximately 60% of AKI patients in clinical practice experience delirium. Elevated creatinine levels>2mg/dL are one of the risk factors for ICU delirium in elderly patients. Renal replacement therapy can reduce the risk of AKI related delirium. For patients receiving renal replacement therapy, daily peak serum creatinine is not related to delirium, but may reduce the impact of AKI on the brain by clearing neurotoxic metabolites. This suggests that renal function has a significant impact on cognitive function in patients, and the gradual normalization of renal function may improve delirium.

Although the underlying mechanism associated with acute renal injury and delirium is still unclear, it has become a consensus that it increases incidence rate and mortality, prolongs hospital stay, and accelerates long-term cognitive decline . The pathogenesis of AKI related delirium is multifactorial, and several hypotheses have been proposed regarding the pathogenesis of AKI induced delirium, including the hypothesis of accumulation of neurotoxins or delirium inducing drugs due to impaired renal clearance function, the hypothesis of upregulation of systemic cytokine mediated neuroinflammatory processes, and the hypothesis of volume overload leading to brain edema.

Multiple studies have identified AKI as the main risk factor for delirium. In a prospective study of 1487 patients, Zipser et al. found that AKI increased the risk of delirium tenfold. A large amount of clinical evidence indicates that the risk of delirium in AKI patients significantly increases with the deterioration of renal function. A retrospective study of 919 ICU patients reported that the incidence of delirium in KDIGO stages 2 and 3 was 20% higher than that in KDIGO stage 1. The BRAIN-ICU study found that 50% of patients have coexisting delirium and AKI. KDIGO stage 2 patients have a 1.5-fold increased risk of delirium, while KDIGO stage 1 patients have a 2.5-fold increased risk of delirium. However, there is no significant correlation between KDIGO stage 1 and delirium. A single center case-control study in the UK further elucidated the role of AKI in different subtypes of delirium. The study showed that KDIGO stage 3 AKI patients were five times more likely to experience excitatory delirium than non AKI patients, and lighter AKI stages (KDIGO stage 1 or 2) were not associated with excitatory delirium.

The above multiple pieces of evidence indicate a significant correlation between AKI and delirium, and both have caused significant losses and burdens to patients and healthcare finances. Given the existence of the renal brain axis and the potential association between AKI and delirium, the investigators hypothesize that by comparing the serum metabolic profiles of patients with delirium and AKI after cardiac surgery, those with only delirium, those with only AKI, and those without delirium and AKI after surgery, the investigators can explore the mechanisms of complications and the interaction mechanisms between organ damage after extracorporeal circulation cardiac surgery, and identify metabolic markers specific to complications, identify patients with increased susceptibility, and provide reference for early diagnosis of complications and basis for early intervention.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old and above
2. Patients undergone elective cardiac surgery
3. History of serum creatinine test within 7 days before surgery
4. Provide venous blood samples
5. Voluntarily participate and sign an informed consent form

Exclusion Criteria:

1. Patients treated with chronic peritoneum or hemodialysis, prior kidney transplantation, preoperative serum creatinine level>4.5mg/dL (400 μ mol/L) or end-stage renal disease (defined as glomerular filtration rate<15ml · min-1 · 1.73m-2)
2. Other related diseases that have been previously confirmed to have cognitive impairment, or records of using drugs targeting cognitive impairment during the onset period
3. Individuals with severe speech, visual, hearing, or mental impairments that affect cognitive scale assessment
4. Individuals with a history of brain tumors, traumatic brain injury, brain parasitic diseases, and other diseases that may cause cognitive impairment
5. Individuals with a history of alcohol and drug addiction
6. Pregnant and lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergone extracorporeal circulation cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2024-07-20 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Small molecule metabolites specific to complications after extracorporeal circulation cardiac surgery | 1 week
  Non biased detection of all small molecule metabolites associated with complications after extracorporeal circulation cardiac surgery, and screening of differential metabolites

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Liu M, Liang Y, Chigurupati S, Lathia JD, Pletnikov M, Sun Z, Crow M, Ross CA, Mattson MP, Rabb H. Acute kidney injury leads to inflammation and functional changes in the brain. J Am Soc Nephrol. 2008 Jul;19(7):1360-70. doi: 10.1681/ASN.2007080901. Epub 2008 Apr 2. PMID 18385426